CLINICAL TRIAL: NCT01213706
Title: Effect of Whole Body Periodic Acceleration on Airway Endothelial Function in Healthy Smokers, Non-smokers and Asthmatics
Brief Title: Effect of Whole Body Periodic Acceleration on Airway Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090748
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Healthy; Smokers; Asthma
Keywords: airway blood flow; albuterol; Whole Body Periodic Acceleration (WBPA); Nitric Oxide; Endothelial Dysfunction
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Body Periodic Acceleration (WBPA) (Experimental): All subjects will be performing this procedure. WBPA in spinal axis (pGz) will be administered with a platform that resembles a bed. The platform moves in a repetitive head-to-foot direction at 140 times a minute, producing 0.22 g.
  Interventions: Device: Whole Body Periodic Acceleration (WBPA); Device: Sham WBPA
- Sham WBPA (Experimental): Sham WBPA :
  All subjects will be performing this procedure before the WBPA. The subjects will rest for 45 minutes in the Whole Body Periodic Acceleration (WBPA) platform without movement as a control challenge.
  Interventions: Device: Whole Body Periodic Acceleration (WBPA); Device: Sham WBPA

INTERVENTIONS:
Device: Whole Body Periodic Acceleration (WBPA) — Subjects will undergo to the Whole Body Periodic Acceleration platform for treatment (shaking period) for 45 min.
Device: Sham WBPA — The subjects will rest for 45 minutes in the Whole Body Periodic Acceleration (WBPA) platform without movement as a control challenge.

SUMMARY:
In the present proposal the investigators wish to assess the effect of a single session with the device known as Exer-Rest® which applies Whole Body Periodic Acceleration (WBPA) on baseline airway blood flow (Qaw) and in Qaw variation, in current smokers, glucocorticoid-naïve asthmatics, and age-matched healthy never-smokers, with the expectation that the treatment will transiently increase the Qaw, and to a greater extent in the current smokers and patients with asthma who have endothelial dysfunction.

DETAILED DESCRIPTION:
Endothelial shear stress activates nitric oxide synthase (NOS), leading to endothelium-dependent vasodilation. This can be accomplished through exercise or with a device known as Exer-Rest® which applies Whole Body Periodic Acceleration (WBPA) that is also called pGz. WBPA produces systemic vasodilation, by exerting shear stress on the vascular endothelium, activating endothelial NOS and releasing NO in animal models and human subjects. Cigarette smoking is associated with attenuated vascular relaxation responses in the systemic circulation. Patients with asthma also exhibit endothelial dysfunction in the airway. In this study the investigators wish to assess the effect of a single pGz session on baseline Qaw and delta Qaw in current smokers, glucocorticoid-naïve asthmatics, and age-matched healthy never-smokers to test if this treatment will increase the vascular relaxation responses.

ELIGIBILITY:
Inclusion Criteria:

15 healthy never-smokers, 15 smokers (> than 1 year smoke history) and 15 never-smokers asthmatics; FEV1 > 80% (except for asthmatics subjets)

Exclusion Criteria:

Women of childbearing potential who do not accepted birth control measures; pregnant and breast feeding; cardiovascular disease or use of cardiovascular drugs; respiratory infection during the 4 weeks preceding the study; use of inhaled or systemic glucocorticoids, leukotriene modifiers or theophyllines in asthmatics; FEV1 < 80% on the screening day (excepted for asthmatics subjets)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- Pulmonary Human Research Laboratory, University of Miami Miller School of Medicine, Miami, Florida, United States

REFERENCES:
- [Background] Sackner MA, Gummels E, Adams JA. Nitric oxide is released into circulation with whole-body, periodic acceleration. Chest. 2005 Jan;127(1):30-9. doi: 10.1378/chest.127.1.30. PMID 15653959
- [Background] Sackner MA, Gummels E, Adams JA. Effect of moderate-intensity exercise, whole-body periodic acceleration, and passive cycling on nitric oxide release into circulation. Chest. 2005 Oct;128(4):2794-803. doi: 10.1378/chest.128.4.2794. PMID 16236957
- [Background] Matsumoto T, Fujita M, Tarutani Y, Yamane T, Takashima H, Nakae I, Horie M. Whole-body periodic acceleration enhances brachial endothelial function. Circ J. 2008 Jan;72(1):139-43. doi: 10.1253/circj.72.139. PMID 18159115

RESULTS

PARTICIPANT FLOW:
Period: Sham WBPA
Arm/Group | SHAM WBPA Then WBPA
Started | 45
Completed | 45
Not Completed | 0
Period: Washout (1 Hour)
Arm/Group | SHAM WBPA Then WBPA
Started | 45
Completed | 45
Not Completed | 0
Period: WBPA
Arm/Group | SHAM WBPA Then WBPA
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Whole Body Periodic Acceleration (WBPA): Whole Body Periodic Acceleration (WBPA) in spinal axis (pGz) will be administered with a platform that resembles a bed. The platform moves in a repetitive head-to-foot direction at 140 times a minute, producing 0.22 g. These settings have been shown to release NO into the circulation.
  Whole Body Periodic Acceleration (WBPA): Subjects will undergo to the Whole Body Periodic Acceleration platform for treatment (shaking period) for 45 min.
Arm/Group | Whole Body Periodic Acceleration (WBPA)
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Airway Blood Flow Response to Albuterol
Description: Airway Blood Flow will be measured before and 15 minutes after the 180 mcg of albuterol inhalation.
Time Frame: Qaw post minus Qaw pre albuterol after WBPA or Sham WBPA
Population: controls n =15, smokers N=15 , asthma N=15
Measure: Mean (Standard Error); unit: μl/min/ml
Groups:
- WBPA: Subjects will undergo to the Whole Body Periodic Acceleration platform for treatment (shaking period) for 45 min.
- Sham WBPA: Subjects will be resting on the platform without any WBPA.
Arm/Group | WBPA | Sham WBPA
Number analyzed (Participants) | 45 | 45
μl/min/ml
  Smokers n=15,15 | 2.85 (2.33) | -1.43 (2.8)
  Controls N=15, 15 | 17.93 (2.08) | 4.03 (0.8)
  Asthma N=15,15 | 1.96 (2.06) | 1.65 (0.8)

ADVERSE EVENTS:
Arm/Group | Whole Body Periodic Acceleration (WBPA) | Sham WBPA
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No